CLINICAL TRIAL: NCT01771081
Title: POLARIS: A Non-interventional Study in Patients With Diabetic Macular Edema (DME) With Central Involvement to Assess the Effectiveness of Existing Anti-vascular Endothelial Growth Factor (Anti-VEGF) Treatment Regimens
Brief Title: Evaluation of Changes in Visual Acuity in Patients With Diabetic Macular Edema (DME) Starting Treatment With an Approved Anti-VEGF Therapy
Acronym: POLARIS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 16459; NN1201 (Other: Company internal)
Record Dates: First submitted 2013-01-11; First posted 2013-01-18 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Ophthalmology; Macular Edema; Macular Degeneration
Keywords: Longitudinal Studies,; Observation; Epidemiology
MeSH Terms: conditions — Macular Edema; Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group1
  Interventions: Drug: Ranibizumab (or other DME treatment)

INTERVENTIONS:
Drug: Ranibizumab (or other DME treatment) — Patients with DME having started treatment with an approved anti-VEGF therapy at or after 01 October 2012 and then continuing with this or any kind or no treatment

SUMMARY:
POLARIS : A non-interventional study in patients with diabetic macular edema (DME) with central involvement to assess the effectiveness of existing anti-vascular endothelial growth factor (anti-VEGF) treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 1 or 2 diabetes mellitus
* Patients diagnosed with DME with central involvement (defined as the area of the center subfield of optical coherence tomography [OCT])
* Patients for whom the decision has been made to treat with an approved anti-VEGF therapy prior to inclusion into the study
* Patients who received the first approved intravitreal anti VEGF treatment from October 01, 2012
* Patients who give informed consent in writing for study participation

Exclusion Criteria:

* Treatment with any anti-VEGF therapy prior to the start of the observation period (October 01, 2012) or enrolment into the study
* Participation in an investigational program with interventions out of clinical routine practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In- and outpatients at participating sites with a diagnosis of DME with central involvement. Patients will be enrolled after the decision for treatment with an approved anti-VEGF therapy has been made at or after October 2012 by the study physician.
Sampling Method: Probability Sample
Enrollment: 911 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in visual acuity, assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) or SNELLEN | Baseline, after 12 months

SECONDARY OUTCOMES:
Demographic and clinical characteristics (Age, sex, race, employment status, severity of DME) | Baseline
Mean time from diagnosis to first commencement with an approved anti-VEGF therapy | Date of first diagnosis; Date of treatment initiation: up to 24 month
Changes in retinal thickness, measured by Optical Coherence Tomography (OCT) | Baseline, after 12 month
Presence of clinically significant macular edema, measured as defined by the ETDRS Research Group | Baseline, after each month, up to 12 month
Resource utilization in terms of treatment choices, frequency and duration | Baseline, after 6 and 12 months
Mean change in quality of life score (using the NEI VFQ 25), only in countries where used as part of routine practice | Baseline, after 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- Many Locations, France
- Many Locations, Germany
- Many Locations, Greece
- Many Locations, Portugal
- Many Locations, Russia
- Many Locations, Slovakia
- Many Locations, Spain
- Many Locations, United Kingdom